CLINICAL TRIAL: NCT03465124
Title: Evaluation of Central Macular Thickness in Femtosecond Laser-assisted Cataract Surgery - FLAME
Brief Title: Evaluation of Central Macular Thickness in Femtosecond Laser-assisted Cataract Surgery
Acronym: FLAME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Menapace, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 1053/2018
Record Dates: First submitted 2018-03-01; First posted 2018-03-14 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Age Related Cataracts; Cystoid Macular Edema
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Intervention Model Description: Bilateral cataract surgery will be performed in individuals with age-related cataract. Eyes will be randomized into two groups receiving either Femtosecond Laser assisted Cataract Surgery (LCS) or conventional Manual Cataract Surgery (MCS).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Groups will be randomized. Randomization information will be put in a sealed envelope on screening date and opened in operating theatre right before procedure start.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femtosecond Laser assisted Cataract Surgery (Active Comparator): Femtosecond Laser assisted Cataract Surgery will be performed unilateral in randomized order.
  Interventions: Device: Femtosecond Laser
- Manual Cataract Surgery (Active Comparator): Manual Cataract Surgery will be performed in contralateral (to LCS) eye of patient with bilateral age-related cataract.
  Interventions: Other: Manual Cataract Surgery

INTERVENTIONS:
Device: Femtosecond Laser — Femtosecond Laser assisted Cataract Surgery will be performed unilateral in randomized order. Contralateral eye will receive conventional cataract surgery
  Arms: Femtosecond Laser assisted Cataract Surgery
Other: Manual Cataract Surgery — conventional cataract surgery as control
  Arms: Manual Cataract Surgery

SUMMARY:
The investigational device is an approved femtosecond laser (FSL) device with an integrated imaging system to perform certain steps of the cataract procedure. The FSL will perform anterior capsulotomy and lens fragmentation in individuals suffering from age-related cataract with need of cataract surgery.

Cataract surgery will be performed in subjects who have signed an informed consent form. Macula thickness will be measured with Spectralis OCT on screening date.

Postoperative examinations will be implemented in accordance with the approved investigational plan on subjects and includes: visual acuity, slitlamp examination, retinal oct imaging and quantitative autofluorescence.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral Age-related cataract necessitating lens extraction and posterior IOL implantation
* Age 40 and older (females of childbearing age will be interviewed if pregnancy is possible)

Exclusion Criteria:

* Corneal abnormality
* Preceding ocular surgery or trauma
* Uncontrolled glaucoma
* Proliferative diabetic retinopathy
* Macular degeneration
* Iris neovascularization
* History of uveitis/iritis
* Microphthalmus
* Recurrent intraocular inflammation of unknown etiology
* Blind fellow eye
* Uncontrolled systemic or ocular disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-04-06 (Estimated)

PRIMARY OUTCOMES:
Central Macular Thickness | Baseline to 6 weeks postoperative
  Difference in Central Macular Thickness (CMT) between Femtosecond Laser-assisted Cataract Surgery (LCS) to Manual Cataract Surgery (MCS)

SECONDARY OUTCOMES:
Influence of lens density on quantitative autofluorescence | Baseline to 1 weel, 3 weeks and 6 weeks postoperative
  Influence of lens density on quantitative autofluorescence will be assessed in qAF units. Images will be recorded after volume scans for each eye on designated visits.
  Quantitative Autofluorescence quantifies natural fundus autofluorescence with a Spectralis HRA+OCT. This method uses the same wavelength and confocal scanning laser ophthalmoscope as fundus autofluorescence (488nm; maximum power: 280 µW) and can be used to determine the integrity and vitality of the retinal pigment epithelium which is important for nourishment the retina.
Central Macular Thickness | Baseline to 1 week, 3 weeks, 6 weeks postoperative
  Difference in Central Macular Thickness (CMT) between Femtosecond Laser-assisted Cataract Surgery (LCS) to Manual Cataract Surgery (MCS)

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Menapace, MD, Principal Investigator — Medical Universitiy of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reiter GS, Schwarzenbacher L, Schartmuller D, Roggla V, Leydolt C, Menapace R, Schmidt-Erfurth U, Sacu S. Influence of lens opacities and cataract severity on quantitative fundus autofluorescence as a secondary outcome of a randomized clinical trial. Sci Rep. 2021 Jun 16;11(1):12685. doi: 10.1038/s41598-021-92309-6. PMID 34135449